CLINICAL TRIAL: NCT02332408
Title: CyberKnife Based Hypofractionated Radiotherapy Versus Conventional Linac Based Radiotherapy for Painful Vertebral Hemangiomas - Controlled Randomized Clinical Trial.
Brief Title: CyberKnife Based Hypofractionated Radiotherapy for Vertebral Hemangiomas
Acronym: CKHRTVH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRVH-COI-03
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Hemangioma of Vertebral Column
Keywords: vertebral hemangioma; conventional radiotherapy; Cyber Knife radiotherapy; randomized trial; radioablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cybernetic microradiosurgery (Experimental): Hypofractionated microradiosurgery using Cyber Knife to the vertebral hemangioma to the total dose of 25 Gy in 5.0 Gy per fraction, 2 or 3 days a week over the period of 2 weeks,
  Interventions: Radiation: Cybernetic microradiosurgery
- Conventional radiotherapy (Active Comparator): Conventionally fractionated external beam conformal radiotherapy to the vertebral hemangioma to the total dose of 36 Gy in 2.0 Gy per fraction, 5 days a week over the period of 3,5 weeks,
  Interventions: Radiation: Conventional radiotherapy

INTERVENTIONS:
Radiation: Cybernetic microradiosurgery — Cybernetic microradiosurgery (6MV) using tracking to TD 25Gy given in five fraction (5Gy p fr) two or three days a week, during 2 weeks
  Arms: Cybernetic microradiosurgery
Radiation: Conventional radiotherapy — Conventionally fractionated linac based external beam radiation therapy - EBRT, (conformal or dynamic) to the TD of 36 Gy, in 2.0 Gy per fraction 5 days a week over the period of 3.5 weeks)
  Arms: Conventional radiotherapy

SUMMARY:
Clinical objective of the study is to compare the analgesic effect, toxicity and pathologic effect in the tumors of two radiotherapy schedules used for patients suffering from painful vertebral haemangiomas

DETAILED DESCRIPTION:
Hemangiomas are frequent vertebral lesions (12% of the whole human population) but only 1% displays any clinical symptoms . The most common symptom is local pain, usually non responding for non-steroid anti-inflammatory drugs. Radiation therapy usually does not result calcification or the tumor regression, but significantly reduces the pain intensity or eliminates it. Currently, the most common RT schedule is conventional radiotherapy using fraction dose (fd) of 2 Gy delivered to the total dose (TD) varying from36 Gy to 40 Gy. The results in pain reduction achieved after larger total doses are better that led us to use radioablative techniques. This procedure is associated with a probability of better analgesic effect and the good local effect (calcification and / or regression of laesion) with high safety of radiation delivery using tracking based cybernetic microradiosurgery (CyberKnife).

The comparison of two modalities of radiation therapy (conventional [fd 2 Gy, TD 36 Gy] and hypofractionated [fd 5 Gy, TD 25 Gy]) used for treatment of painful vertebral hemangioma patients will be performed in the phase III randomized study.

80 patients will be enrolled in this study. All patients will be planned (RT) on the base of CT/MRI fusion.

Patients will be controlled 1, 3, 6, 9, 12 months after treatment completion and, next every each 6 months. Pain relief, analgesics uptake, local effect (MRI and Technetium - 99m-labelled RBC(red blood cell) scintigraphy) and eventual toxicity will be checked during follow-up (FU).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed vertebral hemangioma ,
2. Lesion visible in CT and MR
3. Pain located in area of the lesion
4. Informed consent for participation in the study and for radiotherapy in interested area

Exclusion Criteria:

1. Any previous radiotherapy in region of treated hemangioma
2. Spinal damage or disease that may be associated with an increased radiosensitivity
3. The coexistence of the vertebral morphological changes at the level of hemangioma causing pressure on the nerve roots and / or spinal cord causing pain located in that area
4. Neurological deficits caused by the presence of hemangioma (patients should be considered for surgery)
5. Contradictions for MRI
6. Lack of informed consent.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Analgetic effect | 2 years
  rate of pain relief

SECONDARY OUTCOMES:
Identification of radiologic prognostic and predictal factors of response to external beam radiotherapy (radiosurgery compared to conventional) | 2 years
Identification of biochemical and physical prognostic factors of response to external beam radiotherapy (radiosurgery compared to conventional) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Miszczyk, MD, PhD, Study Director — Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice Branch, Gliwice, Poland
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology Gliwice Branch, Gliwice, Wybrzeze AK 15, Poland

REFERENCES:
- [Background] Sakata K, Hareyama M, Oouchi A, Sido M, Nagakura H, Tamakawa M, Akiba H, Morita K. Radiotherapy of vertebral hemangiomas. Acta Oncol. 1997;36(7):719-24. doi: 10.3109/02841869709001344. PMID 9490090
- [Background] BARTKOWIAK E, BEDNARCZYK J. [CAVERNOUS ANGIOMA OF THE SPINE COMPLICATED BY COMPRESSION VERTEBRAL FRACTURE]. Chir Narzadow Ruchu Ortop Pol. 1964;29:393-6. No abstract available. Polish. PMID 14191260
- [Background] Bremnes RM, Hauge HN, Sagsveen R. Radiotherapy in the treatment of symptomatic vertebral hemangiomas: technical case report. Neurosurgery. 1996 Nov;39(5):1054-8. doi: 10.1097/00006123-199611000-00039. PMID 8905767
- [Background] Heyd R, Seegenschmiedt MH, Rades D, Winkler C, Eich HT, Bruns F, Gosheger G, Willich N, Micke O; German Cooperative Group on Radiotherapy for Benign Diseases. Radiotherapy for symptomatic vertebral hemangiomas: results of a multicenter study and literature review. Int J Radiat Oncol Biol Phys. 2010 May 1;77(1):217-25. doi: 10.1016/j.ijrobp.2009.04.055. Epub 2009 Aug 21. PMID 19699592
- [Background] Asthana AK, Tandon SC, Pant GC, Srivastava A, Pradhan S. Radiation therapy for symptomatic vertebral haemangioma. Clin Oncol (R Coll Radiol). 1990 May;2(3):159-62. doi: 10.1016/s0936-6555(05)80151-7. PMID 2261405
- [Background] Brackrock S, Krull A, Schwarz R, Alberti W. [Results of radiotherapy for vertebral hemangioma]. Strahlenther Onkol. 1999 Aug;175(8):405-8. doi: 10.1007/s000660050029. German. PMID 10481773
- [Background] Faria SL, Schlupp WR, Chiminazzo H Jr. Radiotherapy in the treatment of vertebral hemangiomas. Int J Radiat Oncol Biol Phys. 1985 Feb;11(2):387-90. doi: 10.1016/0360-3016(85)90162-2. PMID 3972655
- [Background] Miszczyk L, Ficek K, Trela K, Spindel J. The efficacy of radiotherapy for vertebral hemangiomas. Neoplasma. 2001;48(1):82-4. PMID 11327544
- [Background] Pavlovitch JM, Nguyen JP, Djindjian M, Mazeron JJ, Piedbois P, Le Bourgeois JP. [Radiotherapy of vertebral hemangioma with neurologic complications]. Neurochirurgie. 1989;35(5):296-8, 305-8. French. PMID 2630926
- [Background] Rades D, Bajrovic A, Alberti W, Rudat V. Is there a dose-effect relationship for the treatment of symptomatic vertebral hemangioma? Int J Radiat Oncol Biol Phys. 2003 Jan 1;55(1):178-81. doi: 10.1016/s0360-3016(02)03734-3. PMID 12504051
- [Background] Schild SE, Buskirk SJ, Frick LM, Cupps RE. Radiotherapy for large symptomatic hemangiomas. Int J Radiat Oncol Biol Phys. 1991 Aug;21(3):729-35. doi: 10.1016/0360-3016(91)90693-x. PMID 1869466
- [Background] Winkler C, Dornfeld S, Baumann M, Christen N, Herrmann T, Eberhardt HJ. [The efficacy of radiotherapy in vertebral hemangiomas]. Strahlenther Onkol. 1996 Dec;172(12):681-4. German. PMID 8992637
- [Background] Yang ZY, Zhang LJ, Chen ZX, Hu HY. Hemangioma of the vertebral column. A report on twenty-three patients with special reference to functional recovery after radiation therapy. Acta Radiol Oncol. 1985 Mar-Apr;24(2):129-32. doi: 10.3109/02841868509134375. PMID 2988274
- [Background] Miszczyk L, Tukiendorf A. Radiotherapy of painful vertebral hemangiomas: the single center retrospective analysis of 137 cases. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):e173-80. doi: 10.1016/j.ijrobp.2011.04.028. Epub 2011 Jun 2. PMID 21640516
- [Background] Gerszten PC, Ozhasoglu C, Burton SA, Vogel WJ, Atkins BA, Kalnicki S, Welch WC. CyberKnife frameless single-fraction stereotactic radiosurgery for benign tumors of the spine. Neurosurg Focus. 2003 May 15;14(5):e16. doi: 10.3171/foc.2003.14.5.17. PMID 15669812
- [Background] Sahgal A, Chou D, Ames C, Ma L, Lamborn K, Huang K, Chuang C, Aiken A, Petti P, Weinstein P, Larson D. Image-guided robotic stereotactic body radiotherapy for benign spinal tumors: theUniversity of California San Francisco preliminary experience. Technol Cancer Res Treat. 2007 Dec;6(6):595-604. doi: 10.1177/153303460700600602. PMID 17994789